CLINICAL TRIAL: NCT03593291
Title: Anti Xa Blood Levels at Survivors of Acute Ischemic Stroke- Receiving LMWH-VTE Prophylaxis
Brief Title: LMWH-VTE Prophylaxis for Survivors of Acute Ischemic Stroke- Assessment of Standard Dosing Regimen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Loewenstein Hospital (Other)
Collaborators: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Motti Ratmansky, MD, PI, Loewenstein Hospital
Other Study IDs: 0022-17-LOE
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: Stroke, VTE prophylaxis, Anti Xa
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anti Xa — Levels of Anti Xa measure

SUMMARY:
The anti-factor Xa (anti-Xa) assay is a functional assay that facilitates the measurement of antithrombin (AT)-catalyzed inhibition of factor Xa by unfractionated heparin (UFH) and direct inhibition of factor Xa by low-molecular-weight heparin (LMWH). As a result, Anti-factor Xa level reflect the in situ pharmacological activity of LMWH. 0.2 to 0.5 units/ml has been considered to be the desired level for prevention of VTE. Although this method was available since the 1970s, their cost was viewed to prohibit their broad use until recently.

Previous studies determined the safety and effectiveness of fixed dose prophylactic regiments via clinical outcomes. This strategy has several shortcomings.

The current study was there for devised to examine in vivo activity of LMWH in patients receiving a fixed dose prophylactic regimen, in order to assess the effectiveness of this method.

DETAILED DESCRIPTION:
The anti-factor Xa (anti-Xa) assay is a functional assay that facilitates the measurement of antithrombin (AT)-catalyzed inhibition of factor Xa by unfractionated heparin (UFH) and direct inhibition of factor Xa by low-molecular-weight heparin (LMWH). As a result, Anti-factor Xa level reflect the in situ pharmacological activity of LMWH. 0.2 to 0.5 units/ml has been considered to be the desired level for prevention of VTE. Although this method was available since the 1970s, their cost was viewed to prohibit their broad use until recently.

Previous studies determined the safety and effectiveness of fixed dose prophylactic regiments via clinical outcomes. This strategy has several shortcomings.

The current study was there for devised to examine in vivo activity of LMWH in patients receiving a fixed dose prophylactic regimen, in order to assess the effectiveness of this method.

Purpose To perform an exploratory prospective analysis of longitudinal data sets to assess anti-factor Xa levels in a cohort of patients recovering from acute ischemic stroke and receiving prophylactic-dose LMWH for VTE prevention.

Primary Outcome Measures:

1. assess anti-factor Xa levels
2. adverse events related to thrombosis
3. adverse event related to hemorrhage

Secondary Outcome Measures:

Patient demographic data Patient anthropometric data Adverse events/weekly (falls, infections, VTE, stress ulcer…) Eligibility

Ages Eligible for Study: 40 Years to 80 Years (Adult, Senior) Gender Eligible for Study: All Accepts Healthy Volunteers: No Sampling Method: Non-Probability Sample Study Population Patients hospitalized for rehabilitation following acute ischemic stroke

Methods:

Clinical decision to administer LMWH prophylactic treatment will be made in line with standard clinical practice and in accordance to the criteria described above.

Search for patients diagnosed with sub-acute stroke and receiving LMWH treatment will be performed on the digital database of the Loewenstien rehabilitation hospital Rannana, Israel.

Patients receiving LMWH prophylaxis with fixed dose regimen will be recruited flowing signing of consent form.

Flowing at least 7 consecutive days of treatment blood sample will be drown 3-4 hours post LMWH administration and sent for The anti-factor Xa (anti-Xa) assay. In the event of high or low results the Hematological consult will be contacted for decision about dose adjustment or other intervention/investigation.

All data will be drawn from patient's electronic/hardcopy files. patient characteristics (age, gender, , past medical history), Stroke characteristics (type, location, NIHSS), days from stroke onset to rehabilitation admission, along with each patient's length of stay, neurological impairments, and Rehabilitation outcomes. Trained research associates, who are familiar with the process of chart review, will extract the information from the charts using the form provided.

Statistical analysis: multi variant combative analysis of outcome measures will be carried out to compare study and control groups.

Estimated Enrollment: 100 patients

ELIGIBILITY:
Inclusion Criteria:

* Acute Ischemic stroke per imaging study
* Clinical decision to administer VTE prophylaxis. (i.e.patients in whom a diagnosis of hemorrhagic stroke has been excluded, the risk of bleeding (hemorrhagic transformation of stroke or bleeding into another site) is assessed to be low, and who have one or more of the following: • major restriction of mobility • previous history of VTE • dehydration or comorbidities (such as malignant disease).Age: 55-80 years)

Exclusion criteria:

* Obese (>150 KG)
* Suffer from renal insufficiency (ccl<30)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for rehabilitation following acute ischemic stroke in 2018
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Anti-Xa level | 3-4 hours post LMWH administration
  Flowing at least 7 consecutive days of treatment blood sample will be drown 3-4 hours post LMWH administration and sent for The anti-factor Xa (anti-Xa) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Motti Ratmansky, MD, Principal Investigator — Loewenstein Hospital
Locations (1):
- Loewenstein Hospital, Raanana, Israel

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available